CLINICAL TRIAL: NCT06677645
Title: Evaluation of Medical and Social Care for Elderly Patients, Between Hospital and Home: TEMPORARY ACCOMMODATION Out of Hospitalization by Nursing Home and Long-Term Care Units in Ile-de-France Region
Acronym: HTSH
Status: Recruiting | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A00023-44
Record Dates: First submitted 2024-10-23; First posted 2024-11-07 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Social Care; Medical Care; Elderly Patients
Keywords: social care; Tempory hospitalization; Elderly people; Medical care; medical-economic study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective group: 258 subjects in the prospective group
- Retrospective group: Retrospective data will be collected directly from hospital departments by ARS IDF or from physicians responsible for medical information (RMI) within each hospital center participating in the study, for the 2 years 2021 and 2022 prior to the study and compared with the average length of stay for services to be calculated at the end of the study.

SUMMARY:
Prospective, observational, non-interventional, comparative, multicenter RIPH3 study to investigate the impact of HTSH on length of hospital stay in referring services.

DETAILED DESCRIPTION:
This is a multi-center study involving many hospital departments temporary accommodation at the end of hospitalization in several Nursing home/long term care units in Ile de France region. The temporary accommodation program was designed for elderly people living at home to find an accommodation solution in nursing home to meet a short-term need. Temporary accommodation beds are deployed and perpetuated in the Île-de-France region by the Regional Health Agency, physically grouped together in establishments within units with dedicated staff. The resources allocated to these beds have been increased. The aim of the study is to demonstrate the efficiency of the HTSH circuit, for elderly patients leaving hospital, in their medical and social care and the decision or not to return home. This project is supported by Regional Health Agency (ARS-IDF).

ELIGIBILITY:
* Inclusion Criteria:

  1. Patient selection criteria

     * Patient male or female at least 60 years of age, as initially defined with the Regional Health Agency, discharged from hospital,
     * Oral expression of non opposition to participation in the study, documented in the medical record by the physician,
     * Presenting a defined and feasible plan for returning home,
     * Whose social/medical situation (stabilized) does not allow an immediate return home after hospitalization.
  2. Caregiver selection criteria

     * Person with an unpaid caregiving activity for their relative in HTSH,
     * Person verbally expressing their non-opposition to participating in the study, and documented in the medical record of the patient they are helping,
     * A person who is able to understand the study questionnaires and evaluations, and is able to answer them without the help of a third party.
  3. Professional selection criteria

     * Salaried professional, nursing or not, regularly and directly involved in the HTSH circuit, whether in hospital or in nursing home / long term care units, for at least 6 months,
     * Oral expression of non opposition to participation in the study, documented by the establishment.
* Non-inclusion Criteria:

  * Be already included in another clinical study,
  * Benefit from a legal protection measure or be unable to express their consent, in accordance with article L1121-8 of the French Public Health Code.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 258 subjects in the prospective group. Retrospective data will be collected directly from hospital departments by ARS IDF or from physicians responsible for medical information (RMI) within each hospital center participating in the study, for the 2 years 2021 and 2022 prior to the study and compared with the average length of stay for services to be calculated at the end of the study.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Study to investigate the impact of HTSH on length of hospital stay in referring services | 24 months
  The main assessment criterion is based on the average length of stay observed at the end of the study, compared with that of the previous two years, 2021 and 2022, in the referring services.

SECONDARY OUTCOMES:
Analysis of pathways and plans for returning home | 24 months
  Evaluation criteria:
  Calculation of the proportion of patients in the life project on admission to nursing home / long term care units and the return home at the end of the stay.
Analysis of HTSH patient profiles a) Proportion of eligible patients and their comorbidities b) Social profile + main reason for hospitalization of patients admitted to HTSH | 24 months
  Evaluation criteria:
  Ratio of hospital ward activity data to pre-screening data collected during the study.
Analysis of discharges and patient outcomes | 24 months
  Proportion of patients remaining at home in the medium term Patients' functional outcome after the trial
Quality of life and caregiver benefit analysis | 24 months
  Quality of life assessment

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Résidence ZEMGOR, Cormeilles-en-Parisis
  - EHPAD Pierre TABANOU, L'Haÿ-les-Roses
  - Groupe Hospitalier Sud Ile de France (GHSIF), Melun
  - GHU Lariboisière, Paris
  - Broca Hospital, Paris
  - USDL Vaugirard, APHP, Paris
  - Centre Hospitalier de Rambouillet, Rambouillet
  - Centre Hospitalier de Versailles, Versailles
  - Hopital Paul Brousse, Villejuif
  - CHU Bicêtre, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code